CLINICAL TRIAL: NCT03635255
Title: Circulating microRNAs and Adverse Cardiovascular Outcomes in Patients With Coronary Artery Disease
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201708063RIND
Record Dates: First submitted 2018-08-15; First posted 2018-08-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: miRNA
Keywords: CAD; miRNA

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood and Urine Sampling After enrollment, 20 mL of blood from peripheral vessels and 10 mL urine were collected. Sampling collection was at the time of enrollment, and every 3 months thereafter in 3-month intervals during outpatient clinic visits. These samples were stored in a -80°C refrigerator until analysis for biomarkers and metabolomic study. Patients were excluded if they had ingested any drugs with antioxidant activity, vitamins, or food additives within the 4 weeks prior to blood/urine sampling.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Coronary artery disease (CAD) resulting from atherosclerotic obstruction of epicardial coronary arteries accounts for more than one-third of deaths in subjects over the age of 35 worldwide. The global incidence of CAD is on the rise owing to the international epidemic of obesity, type 2 diabetes and aging, all of which are potent risk factors for coronary atherosclerosis. Participants with CAD are at high risk for subsequent adverse cardiovascular (CV) events and death; it has been estimated that one out of every five CAD patients will experience at least one adverse CV event during a 5-year follow up period. There is, however, no reliable diagnostic tool to predict the risk of adverse CV events or death in participanrs with CAD. Increasing evidence suggests that miRNAs are stably present in serum, plasma, urine, saliva and other body fluids and are considered a novel class of non-invasive biomarkers for various diseases including cancer, neurodegenerative and cardiovascular diseases

DETAILED DESCRIPTION:
Objective：To identify the novel circulating miRNA expression profiles that may serve as a sensitive and reliable biomarker to predict future adverse CV outcomes and death in patients with established CAD.

Methods：The investigators propose to utilize next-generation sequencing (RNASeq) to identify the novel plasma miRNA expression signature linked to adverse CV outcomes in participanrs with CAD. The identified miRNA candidates that are predictive of adverse CV events will be validated in a larger independent cohort of CAD patients. In addition, miRNAs that are linked to adverse CV outcomes in CAD patients will be investigated mechanistically in human aortic endothelial cells to understand their functional contribution to the occurrence of adverse CV events.

What is New or Innovative in this Study? This study could be one of the few studies to investigate circulating miRNAs as novel biomarkers for risk stratification and the clinical outcome prediction in patients with established CAD. This report will also demonstrate that some dysregulated circulating miRNAs might contribute to endothelial dysfunction and adverse CV events in CAD patients.

Scientific or Clinical Implication of the Expected Results：The results from this study will provide a new prognostic tool to predict CV outcomes in CAD patients using plasma miRNA expression signature. It will also provide important scientific insights into the complex non-coding RNA regulatory network involved in the pathogenesis of atherosclerosis. The insights from this study may provide a unique opportunity to improve the risk assessment of adverse CV events in CAD patients by targeting theses miRNAs.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female older than 20 years old.
2. Have a history of cardiovascular disease (including coronary heart disease, or peripheral vascular disease)

Exclusion Criteria:

Significant valvular or congenital heart disease, cancer, immunosuppressive therapy, or other conditions or treatment your physician thinks you have

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 1. Male or female older than 20 years old.
  2. Have a history of cardiovascular disease (including coronary heart disease, or peripheral vascular disease)
Sampling Method: Probability Sample
Enrollment: 460 (Estimated)
Dates: Start 2019-09-24 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
composite cardiovascular outcome | up to 10 years
  Circulating microRNAs and Adverse Cardiovascular Outcomes in Patients

CONTACTS AND LOCATIONS:
Overall Officials: Chau chung Wu, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- NTUH, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No